CLINICAL TRIAL: NCT05314946
Title: Nutritional Support in Patient Undergoing Induction Therapy for Esophageal Cancer
Brief Title: Nutritional Support During Induction Therapy for Esophageal Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mehdi Qiabi (Other)
Responsible Party: Sponsor-Investigator, Mehdi Qiabi, Associate Scientist, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Organization: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HSREB #120816
Record Dates: First submitted 2022-03-05; First posted 2022-04-07 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Esophageal Cancer; Nutrition Aspect of Cancer
Keywords: cancer; esophagus; enteral nutrition; feeding tube; adverse events; randomized controlled trial; feasibility
MeSH Terms: conditions — Esophageal Neoplasms; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Percutaneous enteral access (Active Comparator): Feeding tube, either gastrostomy (G-) tube or gastrojejunostomy (GJ-) tube (placed by Interventional Radiology) or J-tube (surgically placed)
  Interventions: Procedure: Placement of a percutaneous feeding tube
- No percutaneous enteral access (Experimental): No feeding tube placed.
  Interventions: Procedure: No feeding tube placed

INTERVENTIONS:
Procedure: No feeding tube placed — The experimental arm will forego placement of a feeding tube.
  Arms: No percutaneous enteral access
Procedure: Placement of a percutaneous feeding tube — The standard arm will have a feeding tube placed (G-tube or GJ-tube by IR; or surgically placed J-tube)
  Arms: Percutaneous enteral access

SUMMARY:
Patients diagnosed with esophageal cancer have difficulty eating, as the food pipe becomes obstructed by the cancer. This may impair the ability for the patient to receive appropriate calorie intake, especially during administration of chemotherapy and radiation therapy given prior to surgical resection.

A strategy is to place a feeding tube directly in the stomach or in the small bowel to have an access to the patient's gastrointestinal tract during administration of chemo radiation therapy. However, these feeding tubes may lead to adverse events, including dislodgement, infection, the tube may be plugged, etc. If these complications were to happen, patients may have their treatment delayed, may have to come to the emergency department or even be admitted. In some cases, patients may need to have a surgery performed to treat the complication. Most centres in Canada have moved away from placement of these feeding tubes due to the high incidence of complications associated with the feeding tubes placement, and due to the high efficacy from the chemoradiation therapy in shrinking the tumour, allowing for the patient to swallow.

In London, the preference from the Medical and Radiation Oncologists was to have these feeding tubes placed to avoid delay in treating the patients. There is therefore significant controversy as to what is the best approach in this patient population. Our goal is to run a feasibility randomized controlled trial studying this question.

DETAILED DESCRIPTION:
Esophageal cancer is highly lethal. In Ontario in 2020, an estimated 900 patients were diagnosed with esophageal cancer, while 860 died from it. In Canada, the figures are 2400 diagnoses and 2260 deaths. The incidence of esophageal cancer in Canada is projected to increase over time, especially in males who are more likely to be obese and to suffer from reflux disease.

Esophageal cancer is the malignancy associated with the highest risk for malnutrition. Before their diagnosis, 80% of all patients with esophageal cancer have over 10-15% unintentional weight loss. Strategies to palliate malnutrition in cancer patients and its consequences on outcomes have been developed. In patient with severe nutritional risk, use of nutritional support for at least 10-14 days has been recommended in a non-surgical, oncology population. The European Society for Clinical Nutrition and Metabolism have recommended preoperatively enteral nutrition for 5-7 days in cancer patients undergoing major abdominal surgery. In addition, dietary counselling and oral nutritional supplement were suggested to prevent weight loss and interruption of radiotherapy on patients undergoing radiation treatments for head/neck or gastrointestinal malignancies. Routine enteral nutrition was not suggested during chemotherapy-only treatments.

The type of supplements administered may have an impact on recovery. It was shown that esophageal cancer patients receiving enriched glutamine, fibers and oligosaccharide perioperative enteral supplementation had a shorter systemic inflammatory response syndrome postoperatively and less surgical stress, which could in turn lead to reduced postoperative immunosuppressive conditions. A recent retrospective study from Taiwan did show a slightly improved 4-year overall survival rate and less mucositis on patients supported by enteral feeding tubes with esophageal squamous cell carcinoma and undergoing neoadjuvant therapy.

However, there is still equipoise in the literature and most centers in Canada have moved away from feeding tubes. At LHSC, feeding tubes were historically placed on every patient during their induction treatment. Efforts are being made to spare patients from unnecessary procedure, but patient selection is variable. Standardization of this practice is needed. A recent retrospective study evaluating the effect of surgical enteral access prior to induction treatment did not show nutritional or perioperative benefit. There was no difference in postoperative complication rates and weight loss was similar. In fact, dysphagia is felt to be significantly relieved after a single cycle of chemotherapy. Percutaneous feeding tubes may not be required on all patients during induction therapy for esophageal cancer.

Those feeding tubes are associated with high morbidity. Kidane et al have shown that 39.3% of visits to the ED after an esophagectomy are due to feeding tubes problems (dislodgement, blockage, infection). Of those ED visits for feeding tubes issues, 17% resulted to an admission. Small bowel obstruction is also associated to percutaneous feeding tube placement and selective use has been recommended. Perioperative use of feeding jejunostomy in gastroesophageal cancer has been associate with a complication rate as high as 44%. Given the related-morbidity, guidelines now recommend selective use of feeding tubes on high-risk patients after esophagectomy. When patients undergoing chemotherapy present to the emergency department with fever or infectious signs, data from the Ontario Cancer Registry show that 46% are admitted, increasing healthcare burden. At baseline, patients undergoing chemotherapy are at high risk of presenting to the emergency department or having unplanned visit to the cancer center, this figure going as high as 49% within 4 weeks of initiation of chemotherapy in comparable jurisdictions. Efforts must be made to save an already strained system.

According to the 2020 Surgical Quality Indicator Report Summary from OH-CCO, our center has the worst 30-day unplanned ED visit rate (45%, provincial mean 27%) after esophagectomy in the province of Ontario. Anecdotally, it is felt that most of those cases are related to feeding tubes complications. If these patients present to the ED due to feeding tubes concerns after an esophagectomy, it is likely they would have presented during induction treatment if they had a tube.

Alternative to feeding tubes exist (home IV hydration) which could become a less invasive and more interesting solution.

The objective of this study is to assess the feasibility of a larger randomized controlled trial evaluating unplanned visit to the ED or the outpatient clinic in patients eligible for trimodality for esophageal cancer during their induction treatment, randomized into receiving percutaneous enteral access for nutritional support versus not.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient
* Non-cervical biopsy-proven esophageal or gastroesophageal junction (Siewert I or II) cancer
* Patient eligible for induction therapy then esophagectomy (stage Ib to III)

Exclusion Criteria:

* Impossibility to pass an endoscope beyond the tumour
* metastatic disease
* early-stage disease with either upfront esophagectomy or endoscopic resection planned
* patient refusal of the feeding tube
* inability to swallow their pill
* inability to tolerate a full fluid diet

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility of the trial | From randomization to 90-day post-operative
  The trial will be deemed feasible if 60% or more of eligible patients are recruited, 80% or more of data is collected, and 5% or less patients are lost to follow-up.

SECONDARY OUTCOMES:
Rate of unplanned visits (ED or outpatient clinic) | From randomization to 90-day post-operative
  Rate of unplanned visits (ED or outpatient clinic) from randomization to esophagectomy
Time from PET scan to beginning of induction treatment | From randomization to 90-day post-operative
Total weight loss (kilograms) | From randomization to 90-day post-operative
  Change in kilograms from baseline measured at each visit
Nutritional status | From randomization to 90-day post-operative
  Measured using serum albumin
Any grade adverse event rate | From randomization to 90-day post-operative
Interruption or dose-reduction of the induction treatment | From randomization to 90-day post-operative
Rate of completion of planned induction treatment | From randomization to 90-day post-operative
Quality of life using the Health Related Quality of Life Functional Assessment of Cancer Therapy - Esophageal (HRQOL FACT-E) questionnaire | From randomization to 90-day post-operative
  Higher scores for the scales and subscales indicate better quality of life
Quality of life using the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Oesophago-gastric 25 (EORTC QLQ-OG25) questionnaire | From randomization to 90-day post-operative
  A high score on the functional scales or the global quality of life scale indicates a high function or high level of global quality of life, conversely a high score on a symptom scale represents a high level (severity or frequency, depending on the specific question) of the symptom in question.
Quality of life using the EuroQOL 5 Dimensions 3 Levels (EQ-5D-3L) questionnaire | From randomization to 90-day post-operative
  The maximum score of 1 indicates the best health state, by contrast with the scores of individual questions, where higher scores indicate more severe or frequent problems.
Post-operative morbidity | From surgery to 90-day post-operative
Post-operative mortality | From surgery to 90-day post-operative

CONTACTS AND LOCATIONS:
Locations (1):
- London Health Sciences Centre - Victoria Hospital, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No